CLINICAL TRIAL: NCT01378338
Title: Recurrence Rate, Risk Factors for the Recurrence, and Quality of Life in Patients With GERD in Korea-an Observational Study
Brief Title: Recurrence Rate, Risk Factors for the Recurrence, and Quality of Life in Patients With GERD in Korea-an Observational
Acronym: Refresh
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GKR-ATC-2011/1
Record Dates: First submitted 2011-05-24; First posted 2011-06-22 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: The Aim of This Study is to Investigate the Frequency and Related Risk Factors of Recurrence, and Quality of Life in Patients With GERD After Treatment With PPI
Keywords: GERD; Comparison between ERD and NERD; Rate of complete resolution; rate of recurrence; QOL; To investigate the frequency and related risk factors of recurrence, and quality of life in patients with GERD after treatment with PPI; The aim of this study is to investigate the frequency and related risk factors of recurrence, and quality of life in patients with GERD after treatment with PPI
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Typical reflux symptom by EGD: Total 2000 subjects who has Typical reflux symptom by EGD

SUMMARY:
Recurrence rate, risk factors for the recurrence, and quality of life in patients with GERD in Korea-an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Both ERD or NERD patient who confirmed by EGD findings within 12 months prior to V1 and have a symptom with moderate or more, at least once per week within 1 week prior to V1 and Patients between age 20 and 80with typical reflux symptoms
* Among the patient who have not taken PPI or H2 blocker within 4 weeks prior to V1, needs to be prescribed PPIs 4~8 weeks as a part of the routine clinical practice due to typical symptom
* Patients who give the signed informed consent

Exclusion Criteria:

* Patients with past history of gastrointestinal surgery
* Patients with known malignancy or history of such diseases
* Patients with moderate to severe general medical conditions like ischemic heart disease, chronic renal failure, congestive heart failure, COPD, liver cirrhosis, acute or chronic pancreatitis, or other medical conditions which the investigator considers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with typical reflux symptoms (heartburn or regurgitation) undergone upper endoscopy
Sampling Method: Probability Sample
Enrollment: 855 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence after treatment with PPI in patients with GERD | 12month
Response rate to the treatment with PPI in patients with GERD | 12month

SECONDARY OUTCOMES:
Baseline characteristics related to the recurrence of GERD | 12month
Rate of complete resolution in each group of patients with ERD or NERD | 12month
Rate of recurrence in each group of patients with ERD or NERD | 12month
Quality of life measured by EQ-5D and WPAI-GERD in each group of patients with ERD or NERD | 12month

CONTACTS AND LOCATIONS:
Overall Officials: HyeWon Koo, Study Director — AstraZeneca Korea
Locations (10):
- South Korea (10):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gangneung
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul